CLINICAL TRIAL: NCT03175848
Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Primary Stage IVB Cervical Cancer: A Prospective, Single Arm, Phase II Clinical Trial
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Primary Stage IVB Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-2017-CRT
Record Dates: First submitted 2017-05-28; First posted 2017-06-05 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer Stage IVB
Keywords: Cervical Cancer; Radiotherapy; Chemotherapy; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy,radiotherapy (Experimental): Lymphatic metastasis patients undergoing 2 cycles of chemotherapy(TP/TC), blood metastasis patients receiving 4 cycles of chemotherapy, then patients with therapeutic evaluation for (CR+PR+SD) will undergo the radiotherapy (external irradiation plus brachytherapy) for primary lesion area , all patients completed total 6 cycles of chemotherapy (TP/TC), and finally will determine the of treatment plans of metastasis areas based on tolerance and discuss results by MDT.
  Interventions: Radiation: Chemotherapy,radiotherapy

INTERVENTIONS:
Radiation: Chemotherapy,radiotherapy — Pelvic,pelvic-inguinal,or extended field radiotherapy：Therapy 45 - 50 Gy in 1.7 - 2.0 Gy daily fractions over 4.5 - 5.5 weeks for PTV Brachytherapy: Therapy 5-6 fractions of 4-6Gy prescribed to the high-risk CTV or A piont.

SUMMARY:
This is a prospective, single arm, phase II trail to assess the effect of primary lesion radiotherapy in the treatment of stage IVB cervical cancer on the basis of systemic chemotherapy.

DETAILED DESCRIPTION:
Because of the apparent heterogeneity of stage IVB cervical cancer, at present there is no standard treatment.

This is a Phase II, single-center, single-arm, study of systemic chemotherapy plus lesion radiotherapy for primary stage IVB cervical cancer.

The primary objective of the study is to test the hypothesis that primary lesion radiotherapy leads to an improvement in progression-free survival time (PFS)for stage IVB cervical cancer.

For those patients under the clinical management of the recruiting investigator, the investigator will review the patient's medical records and determine if they would be a candidate for the study.

Upon confirmation of all eligibility criteria, the subject will be enrolled.Patients with beyond abdominal pelvic lymph node metastasis will first undergo 2 cycle systemic chemotherapy（TP/TC），then to evaluate the efficacy of chemotherapy, and for patients with chemotherapy effective（CR+PR+SD) followed by the primary lesion of regional radiotherapy (external irradiation plus brachytherapy)，concurrent chemotherapy （TP/TC） may be given according to the patients tolerant，finally, the patient will complete a total of 6 cycles of chemotherapy（TP/TC）.Distant metastasis of lymph node areas (e.g., supraclavicular, axillary, mediastinum, etc.) will be radiation after radiotherapy at the primary site according to patients tolerant.Patients with stage IVB cervical cancer with hematogenous metastasiswill first undergo 4 cycle systemic chemotherapy（TP/TC），then to evaluate the efficacy of chemotherapy, and for patients with chemotherapy effective（CR+PR+SD) followed by the primary lesion of regional radiotherapy (external irradiation plus brachytherapy)，concurrent chemotherapy （TP/TC） may be given according to the patients tolerant，finally, the patient will complete a total of 6 cycles of chemotherapy（TP/TC），after the primary radiotherapy, the treatment regimen for distant metastasis will be determined by MDT discuss or consultation.Quality of life will be evaluated before and after treatment. During therapy, the patient will have a weekly physical exam, vital signs collected, evaluation for pain, and review any side effects.

Subjects will undergo a post treatment follow-up period after completion of their radiation therapy. During this follow-up period, subjects will return for a medical and history review with a complete physical examination, review of any side effects, evaluation for outcomes and toxicity, and QoL.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven, invasive carcinoma of the cervix(squamous cell carcinoma, adenocarcinoma and adenosquamous carcinoma )
2. KPS≥70
3. FIGO stage IVB
4. Age: 18-70
5. ECOG (Eastern Cooperative Oncology Group) : 0-2
6. The expected survival time is >6 months
7. Chemotherapy and radiation have not been done before
8. Normal hemodynamic indices before the recruitment (including white blood cell count>4.0×109/L, neutrophil count>1.5×109/L, platelet count >100×109/L, hemoglobin≥90g/l, normal liver/kidney function)
9. Able to understand this study and have signed informed consent.

Exclusion Criteria:

1. Prior hysterectomy
2. Metastases lesions are confirmed by pathology or image and are excluded as the second primary neoplasm
3. Patients with brain metastasis or disseminated peritoneal metastasis
4. Female in pregnancy or lactating
5. Hypersensitivity of chemotherapeutic drugs (paclitaxel allergy)
6. History of major psychiatric disorder
7. Persons with physical or mental illness, without civil capacity or with limited capacity for civil conduct
8. Patient with any other disease or condition is a contraindication for chemoradiotherapy
9. The researchers consider the patient not appropriate to be enrolled

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult female cervical cancer patients
Enrollment: 48 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time, PFS | 2 years
  Progression-free survival will be evaluated

SECONDARY OUTCOMES:
Number of Patients with Adverse Events as a Measure of Safety | 2 years
  To quantify rates of acute hematologic, gastrointestinal, and genitourinary toxicity
Objective Response Rates, ORR | 2 years
  Objective Response Rates will be evaluated
Overall survival | 2 years
  Overall survival will be evaluated
Ranking Quality of Life of Patients | 2 years
  To measure health-related quality of life based on the cancer-specific EORTC-QLQ-C30 questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 and cervical cancer module(CX24).
Screening for potentially curable primary stage IVB cervical cancer | 2 years
  By follow-up data,screening for potentially curable primary stage IVB cervical cancer

CONTACTS AND LOCATIONS:
Overall Officials: HanMei Lou, M.A., Principal Investigator — Zhejiang Cancer Hospital; ZhuoMin Yin, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No